CLINICAL TRIAL: NCT05852184
Title: Hb Scope: A Multi-Center Validation Trial
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); SEHA Kidney Care (Unknown); Asia University Hospital (Unknown)
Responsible Party: Principal Investigator, Chin-Chi Kuo, Deputy Superintendent of Big Data Center, China Medical University Hospital
Other Study IDs: T-CMUH-29745
Record Dates: First submitted 2023-03-30; First posted 2023-05-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hemoglobin; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CMUH: Adult patients who receive maintenance hemodialysis through an arteriovenous (AV) fistula or AV graft access at CMUH.
  Interventions: Other: Hb Scope APP
- AUH: Adult patients who receive maintenance hemodialysis through an arteriovenous (AV) fistula or AV graft access at AUH.
  Interventions: Other: Hb Scope APP
- SKC-Central: Adult patients who receive maintenance hemodialysis through an arteriovenous (AV) fistula or AV graft access at SKC-Central.
  Interventions: Other: Hb Scope APP

INTERVENTIONS:
Other: Hb Scope APP — The study intervention is the Hb Scope APP, a camera-based real-time Hb estimation tool using a data collection function and a machine learning-based algorithm to analyze the image of HD tubing and output the estimated Hb value.
  Our proposed Hb Scope APP can provide a non-invasive and real-time estimation of Hb level for detecting the alarming Hb status (i.e., <=10 g/dL) during every HD session. The software is for information management purposes only and is not intended for diagnostic use.

SUMMARY:
The global prevalence of end-stage renal disease (ESRD) was estimated ranging 5.3 to 9.7 million patients in 2017 and is a major healthcare cost driver in both developed and developing economies. The majority of patients with ESRD, approximately 90%, received in-center maintenance hemodialysis (HD). Although HD patients are under the close supervision of a nephrologist, they are vulnerable to anemia and substantial hemoglobin (Hb) variability, which are controversially associated with poor clinical outcomes, such as all-cause mortality. The contemporary narrow target hemoglobin level recommended in the KDIGO and KDOQI guidelines, despite the ongoing debates, poses a crucial challenge in maintaining the optimal hemoglobin level in HD patients.

The Big Data Center at China Medical University Hospital (CMUH) has developed a tool, Hb Scope APP, that can use the color of the HD tubing to predict real-time Hb levels by leveraging the smartphone's camera capacity and machine learning (ML) technology. The performance of the Hb Scope ML algorithm in predicting Hb > 10 g/dL can reach an accuracy of 0.93 and an AUROC of 0.99 in the testing dataset. This opens an opportunity to establish a vibrant digital ecosystem for automatic anemia management.

Innovative ML tools must be appropriately regulated before these algorithms are adopted into clinical practice. Therefore, in the current validation study, we propose to do a multicenter validation trial for validating whether the Hb predicted by Hb Scope APP can achieve an area under the receiver operating curve (AUROC) of at least 0.80 in the adult HD populations from CMUH, Asia University Hospital (AUH) in Taiwan, and SEHA Kidney Care (SKC)-Central in the United Arab Emirates.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving regular maintenance HD in the three participating sites; AND
* Aged 20-90 years old; AND
* Received regular HD through an arteriovenous (AV) fistula or AV graft access; AND
* Use the Fresenius HD machine 4008/4008S and 5008/5008S.

Exclusion Criteria:

* Do not have last Hb level from labs within 1 month prior; OR
* Do not receive blood drawn for the true Hb level or do not have the true Hb level on the date of image taking by Hb Scope APP; OR
* Do not agree to participate.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Study Population: Adult patients receiving regular maintenance HD through an arteriovenous (AV) fistula or AV graft access in the three participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Agreement between the lab-derived and the Hb Scope-derived Hb level at the dichotomous cutoff of > 10 g/dL. | 2 months
  The targeted area under the receiver operating curve (AUROC) is 0.80.

SECONDARY OUTCOMES:
Agreement between the lab-derived and the Hb Scope-derived Hb level at the dichotomous cutoff of < 8 g/dL. | 2 months
  The targeted area under the receiver operating curve (AUROC) is 0.80.
Agreement between the lab-derived and the Hb Scope-derived Hb level at the dichotomous cutoff of > 12 g/dL. | 2 months
  The targeted area under the receiver operating curve (AUROC) is 0.80.
Consistency between the lab-derived and Hb Scope-derived Hb continuous value. | 2 months
  The targeted correlation coefficient is 0.70.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Asia University Hospital, Taichung
- SHEA Kidney Care, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Will not make IPD available to other researchers.